CLINICAL TRIAL: NCT01950143
Title: A Human Dietary Intervention Study to Investigate the Effect of Sulforaphane on Prostate Cancer Interception
Brief Title: Effect of Sulforaphane on Prostate CAncer PrEvention
Acronym: ESCAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Prostate Cancer Foundation (Other); Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IFR01-2013; 14482 (Other: UKCRN)
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2016-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer prevention; diet; global gene expression; metabolic changes
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard broccoli soup (Active Comparator): 26 volunteers
  Interventions: Dietary Supplement: Standard broccoli soup
- Beneforte broccoli soup (Experimental): 26 volunteers
  Interventions: Dietary Supplement: Beneforte broccoli soup
- Beneforte extra broccoli soup (Experimental): 26 volunteers
  Interventions: Dietary Supplement: Beneforte extra broccoli soup

INTERVENTIONS:
Dietary Supplement: Standard broccoli soup — Volunteers will be required to consume one portion of broccoli soup per week as part of their normal diet for one year.
  Arms: Standard broccoli soup
Dietary Supplement: Beneforte broccoli soup — Volunteers will be required to consume one portion per week of a soup containing glucoraphanin-enriched broccoli (Beneforte®) as part of their normal diet for one year.
  Arms: Beneforte broccoli soup
Dietary Supplement: Beneforte extra broccoli soup — Volunteers will be in which they will be required to consume one portion per week of a soup containing an other variety of glucoraphanin-enriched broccoli (Beneforte extra) as part of their normal diet for one year.
  Arms: Beneforte extra broccoli soup

SUMMARY:
The biology of prostate cancer is associated with changes in genes and metabolites within prostate tissue. There is robust evidence to suggest that a diet rich in broccoli can prevent or retard the development of prostate cancer by influencing these changes. This is likely to be due to a natural chemical that is obtained in these vegetables known as sulforaphane.

In this study, we are seeking to provide further evidence that a diet rich in broccoli may prevent prostate cancer from developing, and to understand how this may happen. We propose to undertake a human intervention study to test the hypothesis that a broccoli-rich diet can alter the metabolism and gene expression within prostate tissue of men under active surveillance in a manner that would reduce the probability of the emergence and progression of aggressive cancerous clones. Participants recruited onto this study will be randomly allocated to one of three dietary groups in which they will be required to consume one portion per week of a broccoli soup delivering a different concentration of sulforaphane. This will be part of their normal diet for one year.

Blood, urine and prostate biopsy tissue will be obtained before and after a 12 month intervention period. Prostate biopsies will be obtained either though transperineal template biopsies, a technique accepted as best clinical practice because it provides better sampling of the prostate, or transrectal ultrasound guided biopsy which is currently the standard of care for obtaining biopsies.

This study has been funded by Biotechnology and Biological Sciences Research Council (BBSRC) and Prostate Cancer foundation (PCF).

DETAILED DESCRIPTION:
The study is a randomised double-blinded dietary intervention study. The study population will consist of smoking and non-smoking men aged between 18 and 80 years old. Participants recruited into this study will be randomly placed into one of three dietary groups in which they will be required to consume one portion of broccoli soup per week, delivering a different level of glucoraphanin (sulforaphane precursor), as part of their normal diet for one year. The three types of soup will contain (i)standard broccoli, (ii)glucoraphanin-enriched broccoli (Beneforte®), or (iii)Beneforte extra. Beneforte and Beneforte extra broccoli are especially cultivated to deliver high sulforaphane levels after consumption. All the three broccoli varieties have the same appearance and flavour thus enabling a blinded human intervention study to be undertaken. Broccoli soups will be manufactured by a food company that supplies soups to the leading supermarket retailers in the United Kingdom. In order to assess the habitual diet of the participants, they will be asked to keep three 7-day diet diaries, one pre-intervention, after 6-months and another one week before the end of their intervention. Considering the effect of exercise on whole body metabolism we will also obtain information on the physical activity of study participants. They will be asked to complete a validated physical activity questionnaire together with the diet diary (i.e before starting the study diet then at 6 and 12 months). Twenty six participants will be recruited to each of the broccoli groups. The participants will be characterised as having a low or intermediate risk of developing prostate cancer and will be undergoing active surveillance. A number of physiological tests will be performed on the participants before they start the dietary intervention (baseline) and after their 12 months on the intervention. The study will involve collection of prostate biopsies, blood and urine samples at baseline and after a 12 month dietary intervention. Prostate biopsies will be obtained through transperineal template biopsy (TPB) where possible or standard transrectal ultrasound scan guided biopsy (TRUS biopsy). TPB is a clinical procedure carried out under a general or regional anaesthetic which gives more detailed information about the position, amount and aggressiveness of the cancer within the prostate than other standard techniques. However, patients who do not wish to undergo TPB can alternatively choose the standard TRUS biopsy.

At the end of the trial participants will be asked to give written consent if they wish to continue the diet for a further 12 months. Consenting patients will thereafter be required to eat one portion of broccoli soup per week for 12-months. We will not ask participants to attend extra hospital visits for the purpose of the study or give additional biological samples; instead we will capture clinical data related to their follow up of prostate cancer.

It is anticipated that the dropout rate for this study will be approximately 25% due to the clinical progression of prostate cancer within the 12-month study period. In the event of clinical progression the volunteer will discontinue the intervention, receive advice from the urologist in charge and in case of prostatectomy will be asked to donate part of their prostate gland for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Diagnosed with low and intermediate prostate cancer on active surveillance
* Aged 18-80 years
* BMI between 19.5 and 35 kg/m2
* Smokers and non-smokers

Exclusion Criteria:

* chemopreventive therapy
* 5α-reductase inhibitors or testosterone replacement medicines
* warfarin treatment
* diabetes
* high-risk for human immunodeficiency virus (HIV) and/or hepatitis
* allergy to any of the ingredients of the broccoli soups
* dietary supplements or herbal remedies which may affect the study outcome
* parallel participation in another research project that involves dietary intervention

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-08; Primary Completion 2016-10 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
global gene expression | Baseline and 12 months
  To determine whether a 12 month diet rich in broccoli will result in changes in global gene expression in prostate tissue from men diagnosed with low- and intermediate- risk prostate cancer on active surveillance.

SECONDARY OUTCOMES:
metabolite concentration | Baseline and 12 months
  To determine whether a 12 month diet rich in broccoli will results in changes in levels of metabolites in prostate tissue from men diagnosed with low- and intermediate- risk prostate cancer on active surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Mithen, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Norfolk and Norwich University Hospital, Norwich, United Kingdom

REFERENCES:
- [Derived] Traka MH, Melchini A, Coode-Bate J, Al Kadhi O, Saha S, Defernez M, Troncoso-Rey P, Kibblewhite H, O'Neill CM, Bernuzzi F, Mythen L, Hughes J, Needs PW, Dainty JR, Savva GM, Mills RD, Ball RY, Cooper CS, Mithen RF. Transcriptional changes in prostate of men on active surveillance after a 12-mo glucoraphanin-rich broccoli intervention-results from the Effect of Sulforaphane on prostate CAncer PrEvention (ESCAPE) randomized controlled trial. Am J Clin Nutr. 2019 Apr 1;109(4):1133-1144. doi: 10.1093/ajcn/nqz012. PMID 30982861